CLINICAL TRIAL: NCT03298100
Title: Assessment of Risk Scoring Model for Prediction of Endometrial Cancer Among Symptomatic Postmenopausal Women(a Prospective Cohort Study).
Brief Title: Risk Scoring Model for Endometrial Cancer
Acronym: Cohort
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Asmaa Fahmy Kasem, Assistant lecturer of obestetric and gynecology, Ain Shams University
Other Study IDs: 3176af
Record Dates: First submitted 2017-09-27; First posted 2017-09-29 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postmenopausal women
  Interventions: Other: Scoring model

INTERVENTIONS:
Other: Scoring model — Determining risk factors an calculating the risk score, recurrent vaginal bleeding 3, hypertension 2, age and endometrial thickness 1 for each

SUMMARY:
A prospective cohort study to assess RHEA ( recurrent vaginal bleeding, hypertension, endometrial thickness and age) scoring model for prediction of endometrial carcinoma

ELIGIBILITY:
Inclusion Criteria:

- All postmenopausalwomen with vaginal bleeding and endometrial thickness more than 4 mm

Exclusion Criteria:

* all patients with vaginal bleeding arising from cervical or vaginal or vulval disease or due to hormonal replacement therapy (scheduled bleeding).

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All postmenopausal women (who had their menses stopped for at least one year above age of 40) with vaginal bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-03-20 (Estimated)

PRIMARY OUTCOMES:
Specificity and sensitivity of RHEA scoring mdel | One year
  Positive and negative productive values, specificity and sensitivity of RHEA scoring model

SECONDARY OUTCOMES:
Variables to increase specificity and sensitivity of the score model | One year
  Obesity, diabetes mellitus and family history

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa F Kasem, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided